CLINICAL TRIAL: NCT06336590
Title: Student Exercise and Sleep Timing Study - Part 2
Acronym: SiESTa 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Andrea M. Spaeth, PhD, Primary Investigator, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2024000249
Record Dates: First submitted 2024-02-29; First posted 2024-03-29 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Sleep; Mood; Stress
Keywords: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Exercise (No Intervention): This arm has no intervention. Participants will continue to exercise at their normal evening time (6pm-11pm).
- Morning Exercise (Experimental): Participants will change their exercise times to the morning (6am-11am).
  Interventions: Behavioral: Morning Exercise

INTERVENTIONS:
Behavioral: Morning Exercise — Exercise is changed from normal (6pm-11pm) exercise to morning (6am-11am) exercise.
  Arms: Morning Exercise

SUMMARY:
The purpose of this study is to examine the effects of a morning exercise intervention on sleep (quality and duration), mood (positive affect, anxiety, depression, anger), stress and productivity among undergraduate students (18-23 years) evening-exercisers with poor self-reported sleep quality.

Aim 1. Compared to the control condition, evening-exercisers prescribed morning exercise will exhibit improved sleep quality (increased efficiency, decreased fragmentation) and increased sleep duration.

Aim 2. Compared to the control condition, evening-exercisers prescribed morning exercise will exhibit improved mood (increased positive affect, decreased depression, anxiety and anger).

Aim 3. Compared to the control condition, evening-exercisers prescribed morning exercise will exhibit decreased stress and increased productivity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy undergraduates (18-23 years)
* Frequent evening exercisers (6pm-11pm, 3+ times per week)
* Poor self-reported sleep quality
* Must be willing to wear wrist actigraph 24/7 except when showering/bathing

Exclusion Criteria:

* Sleep/circadian rhythm disorders
* Medications for sleep
* Inability to change schedule to exercise in AM
* Inability to maintain exercise frequency over next 4 weeks

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 2 weeks
  Determine if, compared to a control condition (maintaining usual schedule), shifting exercise from evening to morning improves sleep (quality and duration). Sleep quality includes variables such as the actigraph measured sleep period, total sleep time, sleep efficiency, and wake after sleep onset. Sleep quality and duration will be measured using wrist actigraphy, specifically the Phillips Actiwatch Spectrum Plus devices. The Epworth Sleepiness Scale will also be utilized to measure sleep quality, where scores range from 0-24 and higher scores signify more exhaustion and poorer sleep quality.

SECONDARY OUTCOMES:
Mood | 2 weeks
  Determine if, compared to a control condition (maintaining usual schedule), shifting exercise from evening to morning improves mood (positive affect, depression, anxiety, anger). This will be measure using the Patient-Reported Outcomes Measurement Information System (PROMIS) short form questionnaires for anger, anxiety, depression, and positive affect. Each subsection has a separate score, with higher scores indicating higher levels of anger (scores range from 5-25), anxiety (scores range from 8-40), depression (scores range from 8-40), or positive affect (scores range from 15-75) for each subsection.
Stress | 2 weeks
  Determine if, compared to a control condition (maintaining usual schedule), shifting exercise from evening to morning improves stress levels. This will be measured using the Perceived Stress Scale published in the Journal of Health and Social Behavior in 1983. Higher scores indicate higher stress levels with scores ranging from 0 to 56.
Productivity | 2 weeks
  Determine if, compared to a control condition (maintaining usual schedule), shifting exercise from evening to morning increases productivity. This will be measured using a 5-item questionnaire with a 4-answer scale of poor to excellent (1-4, respectively). The items ask about overall productivity, class attendance, time management, memory, and ability to maintain attention. Higher scores indicate greater productivity with scores ranging from 5 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Spaeth, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (6):
- United States (6):
  - College Avenue Gym, New Brunswick, New Jersey
  - Cook/Douglass Rec Center, New Brunswick, New Jersey
  - Rutgers Fitness Center, New Brunswick, New Jersey
  - Rutgers Sleep Lab, New Brunswick, New Jersey
  - Livingston Rec Center, Piscataway, New Jersey
  - Werblin Rec Center, Piscataway, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
The only IDP sharing that may occur is to other vetted researchers, it will not be made available to all researchers.
Supporting Information: Study Protocol
Time Frame: The deidentified data will be sent to vetted researchers who request it after the data collection period is complete. It will only be available for those vetted researchers for 6 years after the data collection period is complete.